CLINICAL TRIAL: NCT00661180
Title: Open Label Multi-Centric Phase II Study of the Raf Kinase Inhibitor BAY 43-9006 in Chronic Myelogenous Leukemia (CML) Patients Resistant to Gleevec (Imatinib)
Brief Title: Open Label Phase II Study of BAY 43-9006 in Chronic Myelogenous Leukemia (CML) Patients Resistant to Gleevec
Acronym: ORACLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10941; NCT00085007 (obsolete NCT alias)
Expanded Access: Available
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Sorafenib

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Nexavar (Sorafenib, BAY43-9006)

INTERVENTIONS:
Drug: Nexavar (Sorafenib, BAY43-9006) — Patients will receive Bay 43-9006 400 mg po twice daily in a continuous, uninterrupted schedule. Treatment will continue until there is objective evidence of disease progression, or until evidence of toxicities that are unacceptable and thought to be related to study drug, which requires discontinuation of drug, or due to withdrawn patient consent.

SUMMARY:
The purpose of this study is to evaluate the anti-cancer activity and safety of Bay 43-006, in patients who have Chronic Myelogenous Leukemia that resisted to Gleevec treatment, one of the standard medication administered for these patients.

ELIGIBILITY:
Inclusion Criteria:- Have Philadelphia chromosome positive chronic myelogenous leukemia (CML) in chronic phase, as per IBMTR criteria- Have documented hematologic resistance to Gleevec (Imatinib) following a prior hematologic response to Gleevec administered at doses of at least 400 mg/d for at least 3 months.- Have WBC >20 x 109/L at study entry- Have an ECOG performance status. Status of 0, 1 or 2- Have an anticipated survival of at least 16 weeks.- Be able to comply with study procedures and follow-up examinations.- Signed informed consent must be obtained prior to any study specific procedures. Exclusion Criteria:- Congestive heart failure > class II as defined by the New York Heart Association Functional Classification (NYHA)- Cardiac arrhythmias requiring antiarrythmics (excluding beta blockers or digoxin)- Active coronary artery disease or ischemia- History of HIV infection or chronic hepatitis B or C - Active clinically serious infections (> grade 2 NCI-CTC)- Patients with seizure disorder requiring anti-epileptic drugs- History of solid organ allograft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-01; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
To determine the major hematologic response rate (i.e. complete and partial hematologic responses) associated with BAY 43-9006 in patients with chronic phase CML resistant to Gleevec. | Every 3 months

SECONDARY OUTCOMES:
To determine the cytogenetic response rate associated with BAY 43-9006. | Every 3 months
To evaluate the duration of hematologic response to BAY 43-9006. | Throughout study until end of response
To evaluate the duration of cytogenetic response to BAY 43-9006. | Throughout study until end of response
To assess time to progression. | Until event occurs
To assess overall survival.. | During Follow up
To evaluate the molecular response and to perform the pharmacodynamic assessment by analysis the following biomarkers: phospho-Erk, Crkl, phospho-S6 | At 2 months and at last visit
To assess the safety of BAY 43-9006 in patients with chronic phase CML resistant to Gleevec. | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- Portland, Oregon, United States
- France (3):
  - Lyon
  - Paris
  - Poitiers